CLINICAL TRIAL: NCT06732648
Title: The Efficacy and Safety of Intravenous HRS8179 for the Prevention and Treatment of Severe Cerebral Edema Following Large Hemispheric Infarction: a Multicenter, Randomized, Double-blind, Placebo-controlled, Phase II/III Clinical Trial
Brief Title: The Efficacy and Safety of HRS8179 in Severe Cerebral Edema Following Large Hemispheric Infarction
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Beijing Suncadia Pharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HRS8179-301
Record Dates: First submitted 2024-12-10; First posted 2024-12-13 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2024-12

CONDITIONS: Severe Cerebral Edema Following Large Hemispheric Infarction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment group A: HRS8179 injection (Experimental)
  Interventions: Drug: HRS8179 injection
- Treatment group B: HRS8179 injection (Experimental)
  Interventions: Drug: HRS8179 injection
- Treatment group C: HRS8179 blank preparation. (Placebo Comparator)
  Interventions: Drug: HRS8179 blank preparation.

INTERVENTIONS:
Drug: HRS8179 injection — HRS8179 injection; high dose
  Arms: Treatment group A: HRS8179 injection; Treatment group B: HRS8179 injection
Drug: HRS8179 blank preparation. — HRS8179 blank preparation.
  Arms: Treatment group C: HRS8179 blank preparation.

SUMMARY:
The study is being conducted to evaluate the efficacy, and safety of HRS8179 injection in preventing and treating severe cerebral edema after large area cerebral infarction in the cerebral hemisphere

ELIGIBILITY:
Inclusion Criteria:

1. Fully understand and voluntarily participate in this trial, and sign the informed consent form (the informed consent form can be signed voluntarily by the participant or their legal representative);
2. A clinical diagnosis of acute ischemic stroke in the middle cerebral artery (MCA) territory;
3. National Institutes of Health Stroke Scale (NIHSS) ≥ 10 at screening;
4. A large hemispheric infarction defined as: lesion volume of 80 to 160 cm3 on magnetic resonance imaging (MRI) diffusion-weighted imaging (DWI), or computed tomography perfusion (CTP).
5. The time from onset to treatment must be ≤ 10 hours; if the onset time is unknown, treatment must be initiated within 10 hours after the time last known normal.

Exclusion Criteria:

1. Theparticipant is likely to withdraw the supportive treatment on the first day;
2. There is evidence indicating a concurrent infarction in the contralateral hemisphere sufficiently serious to affect functional outcome.
3. There are clinical signs of brain herniation; CT/MRI indicates a midline shift of >2 mm; CT/MRI indicates cerebral hemorrhage;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 725 (Estimated)
Dates: Start 2025-02-07 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Mortality rate at Day 90 | at Day 90

SECONDARY OUTCOMES:
The modified Rankin Scale (mRS) score at Day 90 | at Day 90
The proportion of participants who achieved mRS score 0-4 at Day 90 | at Day 90
Changes in midline shift from baseline to 72 hours | from baseline to 72 hours
The proportion of participants who meet the indications for decompressive craniectomy by Day 14 | Day 14

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided